CLINICAL TRIAL: NCT03955224
Title: Evaluation of Low-Level Laser Therapy Efficacy in Pain Management of Grade 2 Oral Mucositis Induced by Radiotherapy or Chemoradiotherapy: a Phase II Randomized Study in Patients With Upper Aerodigestive Tract Cancer
Brief Title: Evaluation of Low-Level Laser Therapy Efficacy in Pain Management of Grade 2 Oral Mucositis Induced by Radiotherapy or Chemoradiotherapy: a Study in Patients With Upper Aerodigestive Tract Cancer
Acronym: ESMULLLAT
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn due to lack of recruitment
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19 VADS 04
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Upper Aerodigestive Tract Neoplasms
Keywords: Upper Aerodigestive Tract Neoplasms; Low-Level Laser Therapy (LLLT); Mucositis
MeSH Terms: conditions — Head and Neck Neoplasms; Mucositis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Basic Oral Care + active LLLT (experimental arm) (Active Comparator)
  Interventions: Device: Basic Oral Care + active LLLT
- Basic oral Care + inactive LLLT (control arm) (Placebo Comparator)
  Interventions: Other: Basic oral Care + inactive LLLT
- Basic Oral Care (control arm) (Other)
  Interventions: Other: Basic Oral Care

INTERVENTIONS:
Device: Basic Oral Care + active LLLT — * Compliance with the Basic Oral Care Associated with
  * Active LLLT : 5 applications performed at three days intervals (day 1 to day 13 +/- 1 day)
  Arms: Basic Oral Care + active LLLT (experimental arm)
Other: Basic oral Care + inactive LLLT — * Compliance with the Basic Oral Care Associated with
  * Inactive LLLT : 5 applications performed at three days intervals (day 1 to day 13 +/- 1 day)
  Arms: Basic oral Care + inactive LLLT (control arm)
Other: Basic Oral Care — Compliance with the Basic Oral Care only
  Arms: Basic Oral Care (control arm)

SUMMARY:
Prospective, monocentric, randomized phase II study evaluating Low-Level Laser Therapy (LLLT) as a treatment for the pain due to grade 2 oral mucositis in patients with upper aero-digestive tract cancer treated by radiotherapy or chemoradiotherapy.

Patients with upper aero-digestive tract cancer receiving their first cervicofacial radiotherapy or chemoradiotherapy will be included in this study if they suffer from oral mucositis due to their treatment.

The study procedure will consist in 5 applications of the LLLT that will be performed at three days intervals for a maximum duration of 15 days.

Each patient will be followed until 3 days after the end of the study treatment, for a total duration of the study of 18 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Patients with upper aero-digestive tract cancer receiving a first cervicofacial radiotherapy or chemoradiotherapy
3. Patients with a grade 2 mucositis (according to the NCI CTCAE version 5.0) appearing during treatment.
4. Patients available to perform the LLLT treatment: 5 visits at 3 days intervals
5. Patients must provide written informed consent prior to any study specific procedures.
6. Patients affiliated to a Social Health Insurance in France.

Exclusion Criteria:

1. Patients who have already received a cervicofacial radiotherapy
2. Patients who have already received an induction chemotherapy for their upper aero-digestive tract cancer
3. Patients under targeted therapy for their upper aero-digestive tract cancer
4. Patients under systemic corticotherapy
5. Patients with a non-grade 2 mucositis (according to the NCI CTCAE version 5.0)
6. Patients with ulceration or any other oral mucosa pathology than mucositis
7. Pregnant or breastfeeding women
8. Any psychological, familial, geographical or sociological condition which does not allow to respect the medical follow-up and/or compliance to study procedure
9. Patient who has forfeited his/her freedom by administrative or legal award or who is under legal protection (curatorship and guardianship, protection of justice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who didn't need a dose increase or introduction of new analgesics for mouth pain during the study compared to baseline | 16 days for each patient

SECONDARY OUTCOMES:
Evaluation of the oral mucositis pain intensity with Visual Analog Scale Scores | 16 days for each patient
Quality of Life assessed by the Quality of Life Questionnaire specific to Head and Neck cancer (H&N35) | 16 days for each patient
Frequency of adverse events related to the LLLT using the National Cancer Institute Common Toxicity Criteria for Adverse Effects (NCI CTCAE) version 5.0 | 16 days for each patient

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse, France